CLINICAL TRIAL: NCT03039751
Title: Clinical Development and Proof of Principle Testing of New Regenerative Adenovirus Vascular Endothelial Growth Factor (VEGF-D) Therapy for Cost-effective Treatment of Refractory Angina. A Phase II Randomized, Double-blinded, Placebo-controlled Study (ReGenHeart)
Brief Title: Adenovirus Vascular Endothelial Growth Factor D (AdvVEGF-D) Therapy for Treatment of Refractory Angina Pectoris
Acronym: ReGenHeart
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Queen Mary University of London (Other); University College, London (Other); Medical University of Vienna (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); FinVector Vision Therapies Oy (Unknown); Śląski Uniwersytet Medyczny w Katowicach (Unknown); Rigshospitalet, Denmark (Other); Euram Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH5101111
Record Dates: First submitted 2017-01-03; First posted 2017-02-01 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Refractory Angina Pectoris; Gene Transfer; Coronary Artery Disease
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease | interventions — Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AdvVEGF-D (Experimental): Intramyocardial AdVEGF-D
  Interventions: Drug: AdvVEGF-D
- Control (Placebo Comparator): Intramyocardial placebo (buffer solution without gene)
  Interventions: Drug: Control Rx

INTERVENTIONS:
Drug: AdvVEGF-D — AdvVEGF-D will be injected into 10 sites of the myocardium
  Arms: AdvVEGF-D
Drug: Control Rx — Placebo (buffer solution without gene) will be injected into 10 sites of the myocardium
  Arms: Control

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of catheter mediated endocardial adenovirus-mediated vascular endothelial growth factor-D (AdVEGF-D) regenerative gene transfer in patients with refractory angina to whom revascularisation cannot be performed.

DETAILED DESCRIPTION:
Study overview:

The purpose of the study is to evaluate the safety and efficacy of catheter mediated AdVEGF-D regenerative gene transfer in patients with refractory angina to whom revascularisation cannot be performed.

Primary objectives:

To test the efficacy of the therapy to improve functional capacity using 6 minute walking test after 6 months follow-up and improvement of symptoms assessed by Canadian Cardiovascular Society (CCS) class.

Secondary objectives:

Efficacy of the gene transfer to increase to improve functional capacity using 6 minute walking test and improvement of symptoms assessed by CCS class after 12 months as well as increase in myocardial perfusion assessed 6 months after the gene transfer. In addition, at 6 and 12 months timepoints, the improvement quality of life (QoL), the use of angina pectoris medication, major adverse cardiac events related to coronary artery disease (cardiovascular death, myocardial infarction, stroke, revascularization and hospital admission due to coronary artery disease) or a combined endpoint of the above (Major Adverse Cardiac Events, MACE) will be evaluated.

Study design:

ReGenHeart is a randomized, double-blinded, placebo-controlled multicentre phase II study which will be conducted at 6 centers. The study will evaluate the efficacy and safety of catheter mediated endocardial AdVEGF-D regenerative gene transfer in 180 patients with angina pectoris or equivalent symptom despite optimal medical therapy and who are not suitable candidates for coronary revascularization with coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) (refractory angina patients).

Study population:

180 patients will be recruited from the six centers in 2 years. The patients will be selected for the trial on the basis of medical history, general status, laboratory analyses, coronary angiogram and 6-minute walking test. Patients with CCS 2-3 angina pectoris despite optimal medical therapy and who are not eligible for coronary angioplasty or bypass operation due to diffuse coronary stenosis, small coronary vessels, repeated revascularization or too high risk for operation, will be included.

The number of subjects to be recruited and randomized to the trial will be 180 (2:1 ratio to the treatment and control groups).

Investigational drug product:

First generation replication-deficient AdVEGF-D produced in 293 cells will be injected into ten sites in the endocardium. The dose of 1x1011 vp in a total volume of 2 ml (10 times 0.2 ml) will be used. Control patients will be treated and operated exactly in the same way except that placebo (buffer solution without gene) injection into the myocardium is used.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed
* age > 30 but < 85 years
* significant angina pectoris (CCS 2-3) despite of optimal medication
* significant stenosis (> 60%) in coronary angiography (< 6 months)
* contraindication to CABG or PCI due to diffuse or distal stenosis, chronic total occlusion, vessels with difficult anatomy, stenosis with severe calcifications and stenosis in small vessels (<2.5 mm))
* angina pectoris or equivalent symptoms in the 6-minute walking exercise test
* left ventricle wall > 8 mm detected by transthoracic echocardiography or magnetic resonance imaging (treatment area)

Exclusion Criteria:

* women in fertile age
* diabetes mellitus with severe complications such as diabetic retinopathy or nephropathy
* clinically significant anemia (hemoglobin count < 120 mg/l in male, < 110 mg/l in female; hematocrit < 0.36), leukopenia (b-leukocyte count < 3.0x109/l), leukocytosis (b-leukocyte count > 12.0x109/l) or thrombocytopenia (b-thrombocyte count < 100x109/l)
* renal insufficiency (P-creatinine > 160 mg/l)
* liver insufficiency (P-alanine aminotransferase or P-alkaline phosphatase over 2 x normal)
* haematuria of unknown origin
* severe hypertension (systolic blood pressure > 200 mmHg or diastolic blood pressure > 110 mmHg) or significant hypotension (systolic blood pressure < 90 mmHg)
* significant obesity (Body Mass Index > 35)
* acute infection
* immunosuppressive medication
* significant impairment of left ventricular function (ejection fraction < 25% in echocardiography)
* symptomatic congestive heart failure (New York Heart Association class 3-4)
* haemodynamically significant (grade 3-4/4) aortic or mitral regurgitation or other heart disease needing surgery
* recent (< 6 weeks) acute coronary syndrome or myocardial infarction, PCI or CABG, stroke or transient ischemic attack (TIA)
* current or suspected malignancy

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-10-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Functional capacity at 6 months | 6 months after gene transfer
  Improvement of exercise capacity 6 months after the treatment as measured by 6 minute walking test (walking distance in meters)
Severity of angina pectoris symptoms at 6 months | 6 months after gene transfer
  Relieve of angina symptoms 6 months after the treatment (CCS class)

SECONDARY OUTCOMES:
Functional capacity at 12 months | 12 months after gene transfer
  Improvement of exercise capacity 12 months after the treatment as measured by a 6 minute walking test (walking distance in meters)
Severity of angina pectoris symptoms at 12 months | Time Frame: 12 months after gene transfer
  Relieve of angina symptoms 12 months after the treatment (CCS class)
Myocardial perfusion at 6 months | 6 months after gene transfer
  Improvement of myocardial perfusion (myocardial perfusion reserve, MPR) at 6 months assessed with positron emission tomography (PET) or single-photon emission computed tomography (SPECT)
Quality of Life (EQ-5) at 6 and 12 months | 6 and 12 months after gene transfer
  Improvement of QoL assessed with EQ-5 score with three levels of severity and visual analogue scale (VAS) at 6 and 12 months
Quality of Life (Short-Form Health Survey) at 6 and 12 months | 6 and 12 months after gene transfer
  Improvement of QoL assessed with Short-Form Health Survey (SF-36) score at 6 and 12 months
Quality of Life (Seattle Angina Questionnaire ) at 6 and 12 months | 6 and 12 months after gene transfer
  Improvement of QoL assessed with Seattle Angina Questionnaire score at 6 and 12 months
Angina pectoris medication at 6 and 12 months | 6 and 12 months after gene transfer
  Use of short-acting nitrates to relieve symptoms of angina pectoris at 6 and 12 months (number of oral/sublingual nitrate tablets or nitrate spray inhalations during the preceding 4 weeks).
Adverse cardiac events at 6 and 12 months | 6 and 12 months after gene transfer
  Incidence of cardiovascular death, myocardial infarction, stroke, revascularization or hospital admission due to coronary artery disease and a combined endpoint of Major Adverse Cardiac Events MACE (combined endpoint of cardiovascular death, myocardial infarction, stroke, revascularization or hospital admission due to coronary artery disease) at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Seppo Ylä-Herttuala, Study Director — Kuopio University Hospital
Locations (2):
- Rigshospitalet, Copenhagen, Denmark
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
Data wil be shared to Partners of ReGenHeart Consortium